CLINICAL TRIAL: NCT06273995
Title: Telehealth Behavioral Activation for Teens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Texas (Other)
Responsible Party: Principal Investigator, Eric A Storch, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-54233
Record Dates: First submitted 2024-02-13; First posted 2024-02-23 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Depression; Suicide and Self-harm; Depression in Adolescence; Depression Mild; Depression Moderate; Depression Severe
Keywords: behavioral activation; depression; adolescents
MeSH Terms: conditions — Depression; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Single group, open-label behavioral activation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral Activation (BA) (Experimental): Behavioral activation is one such empirically supported intervention. Derived from cognitive-behavioral therapy, a well-established treatment for depression, behavioral activation uses psychoeducation and skill-building to increase an individual's engagement in valued and enjoyable activities (e.g., socializing with family and friends, exercising, participating in a hobby) in order to improve depressive symptoms
  Interventions: Other: Behavioral Activation

INTERVENTIONS:
Other: Behavioral Activation — All participants will undergo behavioral activation treatment for 8-10 weeks

SUMMARY:
Behavioral activation is one such empirically supported intervention. Derived from cognitive-behavioral therapy, a well-established treatment for depression, behavioral activation uses psychoeducation and skill-building to increase an individual's engagement in valued and enjoyable activities (e.g., socializing with family and friends, exercising, participating in a hobby) in order to improve depressive symptoms. Research has shown that behavioral activation is an effective intervention for depressed youth. Additionally, it has been shown as a promising intervention that can be conducted in a brief, virtual format and can be effectively implemented by both trained clinicians and trained, non-licensed interventionists. This project will provide Behavioral Activation for youth (12-17) experiencing depression or suicidal ideation who are currently enrolled in the Youth Depression Suicide Network study in Texas.

DETAILED DESCRIPTION:
Rates of youth depression and suicide are rising worldwide and present a critical public health problem. Between 2007 and 2018, rates of fatal suicide among U.S. youth and young adults increased by 57.4%, becoming the second leading cause of all deaths for Americans between the ages of 10 and 34 in 2020. Similarly, between 2009 and 2019, rates of past year major depressive episodes among adolescents in the United States increased from 8.1% to 15.8% (roughly 1 in 6). Despite these high rates of suicide and depression, Texas is rated 51st in access to mental healthcare in the United States. As untreated youth depression tends to persist and has been related to poorer functioning in adulthood, there is a need to increase access to empirically supported treatment for depressed adolescents.

Behavioral activation is one such empirically supported intervention. Derived from cognitive-behavioral therapy, a well-established treatment for depression, behavioral activation uses psychoeducation and skill-building to increase an individual's engagement in valued and enjoyable activities (e.g., socializing with family and friends, exercising, participating in a hobby) in order to improve depressive symptoms. Research has shown that behavioral activation is an effective intervention for depressed youth. Additionally, it has been shown as a promising intervention that can be conducted in a brief, virtual format and can be effectively implemented by both trained clinicians and trained, non-licensed interventionists.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be enrolled in the Texas Youth Depression Suicide Research Network (TX-YDSRN) Registry Study;
2. Be between the ages of 12- 18 or currently enrolled in high school;
3. Have a caregiver that is willing to participate in the program;
4. Be able to commit to weekly sessions for eight weeks;
5. Be currently experiencing depressive symptoms;
6. Be able to participate in telehealth services within the state of Texas;
7. Be willing to provide consent/assent (parents/legally authorized representative (LAR)/guardian or young adult participant, aged 18 or older, must be willing to provide consent; youth, aged 12-17, must be willing to provide assent);
8. Be able to read, write and speak English or Spanish sufficiently to understand the study procedures and provide written informed consent to participate in the study;
9. Be willing to dedicate appropriate time to complete scheduled study assessment and measures and attend intervention sessions (both parent/LAR/guardian and youth)
10. Be able to provide a reliable means of contact.

Exclusion Criteria:

1. Have an acute medical or psychological condition(s) that that would, in the judgment of the study medical clinician, make participation difficult or unsafe;
2. Have an acute medical or psychological condition(s) that would result in an inability to accurately complete study requirements (e.g., neurological conditions or significant neurodevelopmental concerns);
3. Have active psychotic or manic symptoms resulting in altered mental status and inability to provide assent or requiring immediate attention and/or higher level of intervention;
4. Have a parent/LAR/guardian who is deemed cognitively unable to provide consent (if youth participant, aged 12-17).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9-modified for adolescents (PHQ-A) | During treatment (every session (week) 1-10)
  Depression; 4-point Likert scale (0= Not at all; 3= Nearly every day), Score range 0-27 (higher scores indicate greater depression severity)
Behavioral Activation for Depression-Short Form (BAD-SF) | During treatment (every session (week) 1-10)
  Behavioral Activation; 6-point Likert scale (0= Not al all; 6= Completely), Score range 0-54 (higher scores indicate higher activation)
Dimensional Anhedonia Rating Scale (DARS) | Baseline (before treatment), post-treatment (session/week 11)
  Anhedonia; 5-point Likert scale (0= Not at all; 4= Very much), Score range 0- 68 (higher scores indicate less anhedonia)

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | Baseline (before treatment), post-treatment (session/week 11)
  Behavioral screening; 3-point Likert scale (0= Not at all; 2= Certainly True), Score range 0-40 (higher scores indicate more difficulties)
Duke Social Support Index (DSSI) | Baseline (before treatment), post-treatment (session/week 11)
  Social Support; Multiple Likert scales ((1 = None; 3= More than 2 people)(1= Hardly ever; 3= Most of the time)), Score range 10 -20 (higher scores indicate a higher level of social support)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anvari MS, Hampton T, Tong MP, Kahn G, Triemstra JD, Magidson JF, Felton JW. Behavioral Activation Disseminated by Non-Mental Health Professionals, Paraprofessionals, and Peers: A Systematic Review. Behav Ther. 2023 May;54(3):524-538. doi: 10.1016/j.beth.2022.12.007. Epub 2022 Dec 23. PMID 37088508
- [Background] Copeland WE, Alaie I, Jonsson U, Shanahan L. Associations of Childhood and Adolescent Depression With Adult Psychiatric and Functional Outcomes. J Am Acad Child Adolesc Psychiatry. 2021 May;60(5):604-611. doi: 10.1016/j.jaac.2020.07.895. Epub 2020 Aug 3. PMID 32758528
- [Background] Curtin SC. State Suicide Rates Among Adolescents and Young Adults Aged 10-24: United States, 2000-2018. Natl Vital Stat Rep. 2020 Sep;69(11):1-10. PMID 33054915
- [Background] Daly M. Prevalence of Depression Among Adolescents in the U.S. From 2009 to 2019: Analysis of Trends by Sex, Race/Ethnicity, and Income. J Adolesc Health. 2022 Mar;70(3):496-499. doi: 10.1016/j.jadohealth.2021.08.026. Epub 2021 Oct 16. PMID 34663534
- [Background] Garnett MF, Curtin SC, Stone DM. Suicide Mortality in the United States, 2000-2020. NCHS Data Brief. 2022 Mar;(433):1-8. PMID 35312475
- [Background] Kanter JW, Manos RC, Bowe WM, Baruch DE, Busch AM, Rusch LC. What is behavioral activation? A review of the empirical literature. Clin Psychol Rev. 2010 Aug;30(6):608-20. doi: 10.1016/j.cpr.2010.04.001. PMID 20677369
- [Background] Lebrun-Harris LA, Ghandour RM, Kogan MD, Warren MD. Five-Year Trends in US Children's Health and Well-being, 2016-2020. JAMA Pediatr. 2022 Jul 1;176(7):e220056. doi: 10.1001/jamapediatrics.2022.0056. Epub 2022 Jul 5. PMID 35285883
- [Background] McCauley E, Gudmundsen G, Schloredt K, Martell C, Rhew I, Hubley S, Dimidjian S. The Adolescent Behavioral Activation Program: Adapting Behavioral Activation as a Treatment for Depression in Adolescence. J Clin Child Adolesc Psychol. 2016;45(3):291-304. doi: 10.1080/15374416.2014.979933. Epub 2015 Jan 20. PMID 25602170
- [Background] Reinert, M, Fritze, D. & Nguyen, T. (2021). "The State of Mental Health in America 2022"
- [Background] Ritschel, L. A., Ramirez, C. L., Cooley, J. L., & Craighead, W. E. (2016). Behavioral activation for major depression in adolescents: Results from a pilot study. Clinical Psychology: Science and Practice, 23, 39-57. https://doi.org/10.1111/cpsp.12140
- [Background] Trombello JM, South C, Sanchez A, Kahalnik F, Kennard BD, Trivedi MH. Two Trajectories of Depressive Symptom Reduction Throughout Behavioral Activation Teletherapy Among Underserved, Ethnically Diverse, Primary Care Patients: A VitalSign6 Report. Behav Ther. 2020 Nov;51(6):958-971. doi: 10.1016/j.beth.2020.01.002. Epub 2020 Jan 11. PMID 33051037
- [Background] Uphoff E, Ekers D, Robertson L, Dawson S, Sanger E, South E, Samaan Z, Richards D, Meader N, Churchill R. Behavioural activation therapy for depression in adults. Cochrane Database Syst Rev. 2020 Jul 6;7(7):CD013305. doi: 10.1002/14651858.CD013305.pub2. PMID 32628293